CLINICAL TRIAL: NCT05453331
Title: Asleep MRI-guided and CT-verified Versus Awake Microelectrode Recording Guided Deep Brain Stimulation of the Subthalamic Nucleus in Parkinson's Disease: A Comparative Effectiveness Trial
Brief Title: Asleep MRI-guided Versus Awake Microelectrode Recording Guided Deep Brain Stimulation in Parkinson's Disease: A Comparative Effectiveness Trial
Acronym: ACCURATE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other); HagaZiekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13795
Record Dates: First submitted 2022-06-27; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Parkinson Disease; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Awake MER-guided surgical procedure under local anesthesia with intraoperative testing: Awake micro-electrode recording-guided surgical procedure under local anesthesia with intraoperative testing
  Interventions: Procedure: bilateral STN deep brain stimulation
- Asleep MRI-guided and CT-verified surgical procedure: Asleep MRI-guided and CT-verified surgical procedure
  Interventions: Procedure: bilateral STN deep brain stimulation

INTERVENTIONS:
Procedure: bilateral STN deep brain stimulation — bilateral deep brain stimulation of the subthalamic nucleus in people with Parkinson's disease

SUMMARY:
Rationale: Bilateral deep brain stimulation (DBS) of the subthalamic nucleus (STN) is a well-accepted treatment for Parkinson's disease (PD). Traditionally, the procedure is performed awake and under local anaesthesia to facilitate intraoperative monitoring via microelectrode recording and test stimulation for exact electrode positioning. Advances in MR imaging allow for clear visualization of the STN and therefore direct targeting. Retrospective series suggest that MRI-guided and image (CT or MRI)-verified STN-DBS under general anaesthesia yields a similar motor outcome and quality of life (QoL) as awake and microelectrode recording-guided surgery with intra-operative clinical testing. MRI-guided and image (CT or MRI)- verified approach potentially has advantages in terms of patient experience and cost-effectiveness. The study proposed here is the first in the world to directly compare both methods.

Objective: To compare bilateral MRI-guided and CT-verified STN-DBS under general anaesthesia to awake microelectrode-guided bilateral STN-DBS with intra-operative clinical testing in terms of motor improvement.

Study design: A multicentre comparative effectiveness trial with a non-inferiority design. Study population: 158 PD people eligible for bilateral STN-DBS (79 in each arm).

Intervention: This study compares two modalities of standard treatment. One arm receives awake microelectrode recording guided bilateral STN-DBS under local anaesthesia with intraoperative clinical testing. The other arm receives MRI-guided and CT-verified bilateral STN-DBS under general anaesthesia.

Main study parameters/endpoints: The primary outcome is the change from baseline to one year in Unified Parkinson's Disease Rating Scale part III (UPDRS III) scores (OFF Medication) versus the postoperative scores (OFF medication and ON stimulation). Secondary objectives include patient experience, quality of life, adverse effects and complications, neuropsychological examination, non-motor symptoms (including psychiatric evaluation), reduction in anti-parkinsonian medication, activities of daily living (ADL) functioning and cost- effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* 30-75 years of age
* Idiopathic Parkinson's disease (according to the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease)
* Disease duration ≥ 4 years
* Hoehn & Yahr ≤ 3 (in best ON-medication condition)
* Despite optimal pharmacological treatment, at least one of the following symptoms:
* Disturbing response fluctuation
* Dyskinesia
* Painful dystonia
* Drug-resistant tremor
* ≥30% improvement of Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III score in a levodopa challenge test, except for tremor dominant PD. This is conform daily clinical practice in all participating centres.
* Written informed consent

Exclusion Criteria:

* Dementia (Montreal Cognitive Assessment ≤ 25)
* Previous neurosurgical procedures for PD
* Structural lesions on brain MRI
* Contra-indications for DBS surgery
* Contra-indications for MRI
* Current depression or history recurrent severe depression
* History of psychosis
* Need for nursing care
* Life expectancy < 2 years

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: poeple with Parkinson's disease eligible for bilateral STN-DBS
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale part III | 12 months
  change from baseline to 1 year in Unified Parkinson's Disease Rating Scale part III (min 0, max. 132; higher score means worse outcome)

SECONDARY OUTCOMES:
reduction in anti-parkinsonian medication | 12 months
  change from baseline to 1 year in levodopa equivalent daily dose (LEDD)
health-related quality of life | 12 months
  change from baseline to 1 year in the 39-item Parkinson's Disease Questionnaire (PDQ-39; min. 0, max. 156; higher score means worse outcome)
Non-motor aspects of experiences of daily living | 12 months
  change from baseline to 1 year in Unified Parkinson's Disease Rating Scale part I (min. 0, max. 52; higher score means worse outcome)
Motor aspects of experiences of daily living measured | 12 months
  change from baseline to 1 year in Unified Parkinson's Disease Rating Scale part II (min. 0, max. 52; higher score means worse outcome)
Motor complications after DBS surgery | 12 months
  change from baseline to 1 year in Unified Parkinson's Disease Rating Scale part IV (min. 0, max. 24; higher score means worse outcome)
Patient experience and satisfaction | during hospitalization and follow up visits at approximately 2 weeks after surgery, 6 and 12 months
  Deep Brain Stimulation Patient Experience Rating Scale (min. 0, max. 224, higher score means better outcome)
Depressive symptoms | 12 months
  change from baseline to 1 year in Beck Depression Inventory-Second Edition (BDI-II; min. 0, max. 63, higher score means worse outcome)
Non-Motor Symptoms | 12 months
  change from baseline to 1 year in Non-Motor Symptoms Assessment Scale (NMSS) for Parkinson's disease (min. 0, max. 360, higher score means worse outcome)
Impulsivity | 12 months
  change from baseline to 1 year in Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease (QUIP; min. 0, max. 112, higher score means worse outcome)
Cognitive impairment | 12 months
  change from baseline to 1 year in Montreal Cognitive Assignment (MoCA; min. 0, max. 30, higher score means better outcome)
Anxiety | 12 months
  change from baseline to 1 year in Parkinson Anxiety Scale (PAS, min. 0, max. 12, higher score means worse outcome)
Autonomic symptoms | 12 months
  change from baseline to 1 year in Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction (SCOPA-AUT, min. 0, max. 69, higher score means worse outcome)
Neuropsychiatric symptoms | 12 months
  change from baseline to 1 year in he Neuropsychiatric Inventory Questionnaire (NPI-Q, min. 0, max. 36, higher score means worse outcome)
Patient's sleepiness | 12 months
  change from baseline to 1 year in the Epworth Sleepiness Scale (ESS; min. 0, max. 24; higher score means worse outcome)
Complications and (serious) adverse effects | 12 months
  measured with a standardized check list
Cost effectiveness | during hospitalization (range 3-5 days, median 4 days)
  measured indirectly by duration of operation and duration of hospitalization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abosch A, Timmermann L, Bartley S, Rietkerk HG, Whiting D, Connolly PJ, Lanctin D, Hariz MI. An international survey of deep brain stimulation procedural steps. Stereotact Funct Neurosurg. 2013;91(1):1-11. doi: 10.1159/000343207. Epub 2012 Nov 13. PMID 23154755
- [Background] Ashkan K, Blomstedt P, Zrinzo L, Tisch S, Yousry T, Limousin-Dowsey P, Hariz MI. Variability of the subthalamic nucleus: the case for direct MRI guided targeting. Br J Neurosurg. 2007 Apr;21(2):197-200. doi: 10.1080/02688690701272240. PMID 17453788
- [Background] Binder DK, Rau GM, Starr PA. Risk factors for hemorrhage during microelectrode-guided deep brain stimulator implantation for movement disorders. Neurosurgery. 2005 Apr;56(4):722-32; discussion 722-32. doi: 10.1227/01.neu.0000156473.57196.7e. PMID 15792511
- [Background] Chaudhuri KR, Martinez-Martin P, Brown RG, Sethi K, Stocchi F, Odin P, Ondo W, Abe K, Macphee G, Macmahon D, Barone P, Rabey M, Forbes A, Breen K, Tluk S, Naidu Y, Olanow W, Williams AJ, Thomas S, Rye D, Tsuboi Y, Hand A, Schapira AH. The metric properties of a novel non-motor symptoms scale for Parkinson's disease: Results from an international pilot study. Mov Disord. 2007 Oct 15;22(13):1901-11. doi: 10.1002/mds.21596. PMID 17674410
- [Background] Chen T, Mirzadeh Z, Chapple KM, Lambert M, Shill HA, Moguel-Cobos G, Troster AI, Dhall R, Ponce FA. Clinical outcomes following awake and asleep deep brain stimulation for Parkinson disease. J Neurosurg. 2018 Mar 16;130(1):109-120. doi: 10.3171/2017.8.JNS17883. Epub 2018 Mar 16. PMID 29547091
- [Background] Chircop C, Dingli N, Aquilina A, Zrinzo L, Aquilina J. MRI-verified "asleep" deep brain stimulation in Malta through cross border collaboration: clinical outcome of the first five years. Br J Neurosurg. 2018 Aug;32(4):365-371. doi: 10.1080/02688697.2018.1478061. Epub 2018 May 26. PMID 29806504
- [Background] Counelis GJ, Simuni T, Forman MS, Jaggi JL, Trojanowski JQ, Baltuch GH. Bilateral subthalamic nucleus deep brain stimulation for advanced PD: correlation of intraoperative MER and postoperative MRI with neuropathological findings. Mov Disord. 2003 Sep;18(9):1062-5. doi: 10.1002/mds.10489. PMID 14502679
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Deuschl G, Schade-Brittinger C, Krack P, Volkmann J, Schafer H, Botzel K, Daniels C, Deutschlander A, Dillmann U, Eisner W, Gruber D, Hamel W, Herzog J, Hilker R, Klebe S, Kloss M, Koy J, Krause M, Kupsch A, Lorenz D, Lorenzl S, Mehdorn HM, Moringlane JR, Oertel W, Pinsker MO, Reichmann H, Reuss A, Schneider GH, Schnitzler A, Steude U, Sturm V, Timmermann L, Tronnier V, Trottenberg T, Wojtecki L, Wolf E, Poewe W, Voges J; German Parkinson Study Group, Neurostimulation Section. A randomized trial of deep-brain stimulation for Parkinson's disease. N Engl J Med. 2006 Aug 31;355(9):896-908. doi: 10.1056/NEJMoa060281. PMID 16943402
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] Ford I, Norrie J. Pragmatic Trials. N Engl J Med. 2016 Aug 4;375(5):454-63. doi: 10.1056/NEJMra1510059. No abstract available. PMID 27518663
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Gorgulho A, De Salles AA, Frighetto L, Behnke E. Incidence of hemorrhage associated with electrophysiological studies performed using macroelectrodes and microelectrodes in functional neurosurgery. J Neurosurg. 2005 May;102(5):888-96. doi: 10.3171/jns.2005.102.5.0888. PMID 15926715
- [Background] Hariz M, Blomstedt P, Limousin P. The myth of microelectrode recording in ensuring a precise location of the DBS electrode within the sensorimotor part of the subthalamic nucleus. Mov Disord. 2004 Jul;19(7):863-864. doi: 10.1002/mds.20135. No abstract available. PMID 15254958
- [Background] Hariz MI, Krack P, Melvill R, Jorgensen JV, Hamel W, Hirabayashi H, Lenders M, Wesslen N, Tengvar M, Yousry TA. A quick and universal method for stereotactic visualization of the subthalamic nucleus before and after implantation of deep brain stimulation electrodes. Stereotact Funct Neurosurg. 2003;80(1-4):96-101. doi: 10.1159/000075167. PMID 14745216
- [Background] Ho AL, Ali R, Connolly ID, Henderson JM, Dhall R, Stein SC, Halpern CH. Awake versus asleep deep brain stimulation for Parkinson's disease: a critical comparison and meta-analysis. J Neurol Neurosurg Psychiatry. 2018 Jul;89(7):687-691. doi: 10.1136/jnnp-2016-314500. Epub 2017 Mar 1. PMID 28250028
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] LaHue SC, Ostrem JL, Galifianakis NB, San Luciano M, Ziman N, Wang S, Racine CA, Starr PA, Larson PS, Katz M. Parkinson's disease patient preference and experience with various methods of DBS lead placement. Parkinsonism Relat Disord. 2017 Aug;41:25-30. doi: 10.1016/j.parkreldis.2017.04.010. Epub 2017 Apr 17. PMID 28615151
- [Background] Leentjens AF, Dujardin K, Pontone GM, Starkstein SE, Weintraub D, Martinez-Martin P. The Parkinson Anxiety Scale (PAS): development and validation of a new anxiety scale. Mov Disord. 2014 Jul;29(8):1035-43. doi: 10.1002/mds.25919. Epub 2014 May 23. PMID 24862344
- [Background] Limousin P, Pollak P, Benazzouz A, Hoffmann D, Le Bas JF, Broussolle E, Perret JE, Benabid AL. Effect of parkinsonian signs and symptoms of bilateral subthalamic nucleus stimulation. Lancet. 1995 Jan 14;345(8942):91-5. doi: 10.1016/s0140-6736(95)90062-4. PMID 7815888
- [Background] Marinus J, Visser M, Jenkinson C, Stiggelbout AM. Evaluation of the Dutch version of the Parkinson's Disease Questionnaire 39. Parkinsonism Relat Disord. 2008;14(1):24-7. doi: 10.1016/j.parkreldis.2007.05.005. Epub 2007 Aug 16. PMID 17702633
- [Background] McClelland S 3rd. A cost analysis of intraoperative microelectrode recording during subthalamic stimulation for Parkinson's disease. Mov Disord. 2011 Jul;26(8):1422-7. doi: 10.1002/mds.23787. Epub 2011 Jun 14. PMID 21674622
- [Background] Nakajima T, Zrinzo L, Foltynie T, Olmos IA, Taylor C, Hariz MI, Limousin P. MRI-guided subthalamic nucleus deep brain stimulation without microelectrode recording: can we dispense with surgery under local anaesthesia? Stereotact Funct Neurosurg. 2011;89(5):318-25. doi: 10.1159/000330379. Epub 2011 Sep 15. PMID 21921673
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Thissen AJ, van Bergen F, de Jonghe JF, Kessels RP, Dautzenberg PL. [Applicability and validity of the Dutch version of the Montreal Cognitive Assessment (moCA-d) in diagnosing MCI]. Tijdschr Gerontol Geriatr. 2010 Dec;41(6):231-40. doi: 10.1007/s12439-010-0218-0. Dutch. PMID 21229776
- [Background] Tomlinson CL, Stowe R, Patel S, Rick C, Gray R, Clarke CE. Systematic review of levodopa dose equivalency reporting in Parkinson's disease. Mov Disord. 2010 Nov 15;25(15):2649-53. doi: 10.1002/mds.23429. PMID 21069833
- [Background] Vinke RS, Selvaraj AK, Geerlings M, Georgiev D, Sadikov A, Kubben PL, Doorduin J, Praamstra P, Bloem BR, Bartels RHMA, Esselink RAJ. The Role of Microelectrode Recording and Stereotactic Computed Tomography in Verifying Lead Placement During Awake MRI-Guided Subthalamic Nucleus Deep Brain Stimulation for Parkinson's Disease. J Parkinsons Dis. 2022;12(4):1269-1278. doi: 10.3233/JPD-223149. PMID 35367970
- [Background] Visser M, Marinus J, Stiggelbout AM, Van Hilten JJ. Assessment of autonomic dysfunction in Parkinson's disease: the SCOPA-AUT. Mov Disord. 2004 Nov;19(11):1306-12. doi: 10.1002/mds.20153. PMID 15390007
- [Background] Weintraub D, Mamikonyan E, Papay K, Shea JA, Xie SX, Siderowf A. Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale. Mov Disord. 2012 Feb;27(2):242-7. doi: 10.1002/mds.24023. Epub 2011 Dec 1. PMID 22134954
- [Background] Wodarg F, Herzog J, Reese R, Falk D, Pinsker MO, Steigerwald F, Jansen O, Deuschl G, Mehdorn HM, Volkmann J. Stimulation site within the MRI-defined STN predicts postoperative motor outcome. Mov Disord. 2012 Jun;27(7):874-9. doi: 10.1002/mds.25006. Epub 2012 Apr 19. PMID 22517070
- [Background] Xiaowu H, Xiufeng J, Xiaoping Z, Bin H, Laixing W, Yiqun C, Jinchuan L, Aiguo J, Jianmin L. Risks of intracranial hemorrhage in patients with Parkinson's disease receiving deep brain stimulation and ablation. Parkinsonism Relat Disord. 2010 Feb;16(2):96-100. doi: 10.1016/j.parkreldis.2009.07.013. Epub 2009 Aug 13. PMID 19682943
- [Background] Zrinzo L, Foltynie T, Limousin P, Hariz MI. Reducing hemorrhagic complications in functional neurosurgery: a large case series and systematic literature review. J Neurosurg. 2012 Jan;116(1):84-94. doi: 10.3171/2011.8.JNS101407. Epub 2011 Sep 9. PMID 21905798